CLINICAL TRIAL: NCT01671163
Title: EUS-Guided Fiducial Placement for Stereotactic Body Radiotherapy
Brief Title: Endoscopic Ultrasound-Guided Fiducial Placement for Stereotactic Body Radiotherapy
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600243; 326-2012 (Other: University of Florida Institutional Review Board)
Record Dates: First submitted 2012-08-01; First posted 2012-08-23 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Cancer
Keywords: Cancer; Radiation therapy; Fiducial markers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects requiring fiducial placement: Endoscopic Ultrasound (EUS) for fiducial placement
  Interventions: Procedure: Endoscopic Ultrasound (EUS) for fiducial placement

INTERVENTIONS:
Procedure: Endoscopic Ultrasound (EUS) for fiducial placement — Endoscopic Ultrasound (EUS) used for the placement of fiducial markers in tissue as outlined by the radiation oncologist

SUMMARY:
The purpose of this research study is to evaluate placing the radiation therapy markers (Fiducial) by using an endoscopic procedure. The endoscopic procedure is called an Endoscopic Ultrasound (EUS). This is a procedure using a special endoscope that has an ultrasound on the end. The ultrasound will allow the doctor's to see where the radiation therapy markers (Fiducial) is to be placed as outlined by the Radiation Oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* Scheduled to undergo fiducial placement,
* Subject must be able to give informed consent

Exclusion Criteria:

* Any contraindication to performing endoscopy,
* Participation in another research protocol that could interfere or influence the outcomes measures of the present study,
* The subject is unable/unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who are currently scheduled to undergo fiducial placement at the University of Florida in Gainesville as medically indicated.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the success and accuracy of endoscopic delivery of the Fiducials into pre-selected targets using dedicated EUS fiducial delivery system. | approximately one week
  The outcome measure for this study is to determine:
  1. The successful delivery, to the targeted tissue,of the fiducials through the fiducial delivery system,
  2. The accuracy of the fiducial delivery into the targeted tissue and
  3. to see if the fiducials can be visualized via Endoscopic Ultrasound (EUS), Fluoroscopy and/or CT scan.
  The success and accuracy of the delivery will be evaluated by Endoscopic Ultrasound, fluoroscopy and/or CT scan to determine if the fiducials are in the targeted tissue. The subject's Oncologist will inform the endoscopist of the targeted tissue that is to receive the fiducials.

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida; Robert Zlotecki, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida/Shands, Gainesville, Florida, United States